CLINICAL TRIAL: NCT04388995
Title: Stroke Volume Variation and Pulse Pressure Variation Predict Fluid Responsiveness in Mechanically Ventilated Elderly Patients Under General Anesthesia
Brief Title: SVV and PPV Predict Fluid Responsiveness in Mechanically Ventilated Elderly Patients Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yi Liu, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PLAGHAOC202002
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Stroke Volume Variation; Pulse Pressure Variation; Fluid Responsiveness; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observed patients (Experimental)
  Interventions: Diagnostic Test: volume expansion

INTERVENTIONS:
Diagnostic Test: volume expansion — volume expansion with 6% hydroxyethyl starch (7 mL/kg) at a rate of 0.4 mL/kg/min

SUMMARY:
Although individualized or goal-directed approach has been advocated, a reliable index is still required to help monitor the volume status timely and efficiently. Dynamic indexes, such as pulse pressure variation (PPV) and stroke volume variation (SVV), have been shown to be clearly superior to more commonly measured static preload variables, such as pulmonary artery occlusion pressure (PAOP) and central venous pressure (CVP). The reliability of dynamic indexes in monitoring the volume status and predicting fluid responsiveness have been validated. Fluid optimization guided by SVV and PPV is beneficial to hemodynamic stability and can decrease mortality and reduce postoperative complications. However, the usefulness of dynamic indexes in elderly patients has not been previously investigated. This study aimed to evaluate whether dynamic indexes PPV and SVV can reliably predict fluid responsiveness in elderly patients, and to determine their thresholds in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients undergoing gastrointestinal surgery 2.Age between 18 and 80 3.ASA I ~II. 4.BMI 18 ~ 24 kg/m2

Exclusion Criteria:

* 1.arrhythmias 2.intracardiac shunts 3.severe hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg) 4.pulmonary hypertension 5.chronic obstructive pulmonary disease 6.peripheral vascular obstructive disease 7.receiving long-term treatment with vasopressors.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | immediately after the fluid therapy
  Fluid responsiveness was defined as an increase in CI ≥15%

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China